CLINICAL TRIAL: NCT05390814
Title: [18F]-Fludarabine PET/MR Imaging for the Assessment of Newly-diagnosed Primary Central Nervous System (CNS) Lymphoma : a Pilot PET-MRI Study
Brief Title: [18F]-Fludarabine PET/MRI in Primary Central Nervous System Lymphoma
Acronym: FLUDALOC
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: P160407; 2021-005193-26 (EudraCT Number)
Record Dates: First submitted 2022-05-20; First posted 2022-05-25 (Actual); Last update posted 2025-08-22 (Actual); Status verified 2025-08

CONDITIONS: Primary Central Nervous System Lymphoma
Keywords: [18F]-Fludarabine; PET-MRI; Primary Central Nervous System Lymphomas

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- PET-RMI (Experimental)
  Interventions: Drug: PET-MRI

INTERVENTIONS:
Drug: PET-MRI — [18F]-Fludarabine imaging in the diagnostic workup of primary central nervous system lymphomas: a PET-MRI pilot study

SUMMARY:
Primary central nervous system (CNS) lymphomas represent 5% of primary brain tumors. More than 90% of them are diffuse large B-cell lymphomas.

[18F]-Fluorodeoxyglucose positron emission tomography (PET-[18F]-FDG) is the gold standard for imaging systemic lymphomas, but its application in primary CNS lymphoma is compromised by the limited specificity of brain fixations and the high uptake of [18F]-FDG in healthy brain tissue.

[18F]-Fludarabine is a new radiopharmaceutical developed for PET imaging of lymphomas. Preclinical studies indicate a restricted binding specificity to lymphoid tissue compared to [18F]-FDG and an ability to detect residual lymphoma disease after treatment. A pilot study in humans shows good agreement of its binding with tumor sites in systemic lymphoma and superior tumor contrast to [18F]-FDG. Finally, a recent preclinical study shows a binding ratio in brain lymphoma 3 times higher than that of healthy brain tissue in mouse models of primary CNS lymphoma, whereas in mouse models of high-grade glial tumors, the binding level is very low, comparable to that of healthy tissue (background). Investigators hypothesize that [18F]-Fludarabine could be the radiopharmaceutical of choice for the diagnosis and monitoring of primary CNS lymphomas in PET.

The main objective of the study is to characterize the cerebral distribution and [18F]-Fludarabine uptake in newly-diagnosed primary CNS lymphomas before surgery, chemotherapy or radiotherapy, using PET-MR imaging.

DETAILED DESCRIPTION:
Monocenter, open, uncontrolled and non-randomized pilot study designed to evaluate the uptake of [18F]-Fludarabine in 16 patients with newly diagnosed CNS lymphoma at initial diagnosis, before treatment using hybrid PET/MR system.

Main objective: to characterize the brain distribution and tumoral uptake in CNS lymphoma before treatment. The secondary objectives are to compare PET-[18F]-Fludarabine results with those of morphological MRI with and without gadolinium injection, diffusion and perfusion MRI, proton-spectroscopy, histological or cytological diagnosis, and brain [18F]-FDG PET imaging.

Patient screening includes a clinical and neurological examination, diagnostic MRI, biological examination, [18F]-FDG PET examination to exclude systemic lymphoma, histological/cytological diagnosis of brain lymphoma. Once informed consent is obtained, one brain PET with [18F]-Fludarabine (4 MBq/kg) combined with simultaneous multiparametric MR sequences is scheduled.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged ≥ 18 years
* Diagnosis of newly diagnosed high-grade CNS lymphoma (with histological and/or cytological confirmation)
* Patient naive to chemotherapy, or radiotherapy treatment for CNS lymphoma
* Contrast-enhanced intracranial mass greater than or equal to 1 cm longest axis
* Karnofsky index ≥ 40
* No systemic lymphoma on [18F]-FDG PET/CT
* Creatinine clearance ≥ 30 mL/min
* Social security affiliation (excluding AME)
* Signature of the informed consent by the patient or by a legal representative or the close relative if the patient is not able to do so

Exclusion Criteria:

* Hypersensitivity to the active substance, to any of the excipients or to any of the components of [18F]-Fludarabine
* Previous treatment for primary central nervous system lymphoma
* Isolated primary vitro-retinal lymphoma
* Isolated CNS relapse of a systemic lymphoma
* Other active cancer except basal cell carcinoma of the skin and/or cervical cancer in situ
* Immunosuppression (organ transplant in particular)
* Positive HIV serology
* Presence of another progressive pathology that is life-threatening in the short term
* Treatment with dipyridamole
* History of allergy to gadolinium chelates (DOTAREM®)
* Absolute contraindication to MRI (pacemaker, cochlear implant ...), to the administration of gadolinium
* Patient of childbearing potential without effective contraception, breastfeeding or pregnant
* Severe cognitive impairment incompatible with good cooperation in the PET-MRI examination
* Patient with pain or restlessness unable to remain motionless in supine position for 60 minutes
* Weight > 100 Kg
* Patient deprived of liberty or under legal protection (guardianship or curatorship)
* Ongoing participation in another interventional research protocol. Participation in research of a non-interventional type is authorized.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2023-12-18 (Actual); Primary Completion 2024-12-05 (Actual); Study Completion 2024-12-05 (Actual)

PRIMARY OUTCOMES:
Measurements of [18F]-Fludarabine uptake in tumoral lesions and normal tissue using SUV, tumor/normal tissues ratios | 15 days
  Standardized measurement of [18F]-Fludarabine uptake (SUV) in tumor will be done on PET imaging superimposed on post gadolinium MRI.

SECONDARY OUTCOMES:
Cerebral distribution of [18F]-Fludarabine in healthy and tumoral tissues | 15 days
  [18F]-Fludarabine time activity curves will be generated in normal and tumoral tissues with dynamic PET acquisition
Temporal activity curves of [18F]-Fludarabine in healthy and tumoral tissues | 15 days
  [18F]-Fludarabine time activity curves will be generated in normal and tumoral tissues with dynamic PET acquisition
Tumor SUVmax, tumor/healthy tissue ratio in PET- [18F]-FDG | 15 days
  Tumoral uptake in [18F]-FDG brain PET and brain [18F]-Fludarabine will be compared as well as contrast to normal uptake
Volumes of contrast enhancement in post-gadolinium T1-weighted MR sequence | 15 days
  Tumor uptake delimitation will be compared to contrast enhancement limits
Hypersignal in diffusion-weighted sequence and apparent diffusion coefficient (ADC) | 15 days
  Tumor volume on brain PET will be compared to hypersignal volume on T2-weighted FLAIR sequence
Tumor perfusion, capillary permeability in perfusion weighted MRI | 15 days
  [18F]-Fludarabine uptake in tumor will be analyzed in light of tumor perfusion on PET superimposed on perfusion sequence
Metabolite ratios in spectroscopy | 15 days
  [18F]-Fludarabine uptake in tumor will be analyzed in light of metabolites profile in proton-spectroscopy

CONTACTS AND LOCATIONS:
Overall Officials: Aurélie KAS, Pr, Principal Investigator — Assistance Publique - Hôpitaux de Paris
Locations (1):
- Hôpital Pitié Salpêtrière, Paris, France

IPD SHARING:
Plan to Share IPD: Yes
The procedures carried out with the French data privacy authority (CNIL, Commission nationale de l'informatique et des libertés) do not provide for the transmission of the database, nor do the information and consent documents signed by the patients. Consultation by the editorial board or interested researchers of individual participant data that underlie the results reported in the article after deidentification may nevertheless be considered, subject to prior determination of the terms and conditions of such consultation and in respect for compliance with the applicable regulations.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Beginning 3 months and ending 3 years following article publication. Requests out of these time frame can also be submitted to the sponsor
Access Criteria: Researchers who provide a methodologically sound proposal.